CLINICAL TRIAL: NCT05276375
Title: Effect of Bronchipret on Antiviral Immune Response in Patients With Mild COVID-19 (BroVID)
Brief Title: Effect of Bronchipret on Antiviral Immune Response in Patients With Mild COVID-19
Acronym: BroVID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Frank Behrens (Other)
Collaborators: Bionorica SE (Industry)
Responsible Party: Sponsor-Investigator, Dr. Frank Behrens, Sponsor representative, Fraunhofer Institute for Translational Medicine and Pharmacology ITMP
Organization: Fraunhofer Institute for Translational Medicine and Pharmacology ITMP (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMP-2005-2020-36
Record Dates: First submitted 2022-03-02; First posted 2022-03-11 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: COVID-19
Keywords: ARDS; COVID 19; Bronchipret
MeSH Terms: conditions — COVID-19 | interventions — thyme extract and ivy extract drug combination

STUDY DESIGN:
Intervention Model Description: Comparison of Verum (Bronchipret) versus no verum i.d. standard of care
Masking Description: open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bronchipret (Active Comparator): Bronchipret syrup (3x 5,4 ml daily, according to summary of product characteristics) until day 14
  Interventions: Drug: Bronchipret
- standard of care (No Intervention): no study intervention

INTERVENTIONS:
Drug: Bronchipret — Bronchipret syrup (3x 5,4 ml daily) until day 14
  Arms: Bronchipret

SUMMARY:
There is currently an urgent need for effective and safe treatments of Coronavirus Disease (COVID) - 19 and the cytokine storm that is responsible for the development of patient's Acute Respiratory Distress Syndrome (ARDS).

As Bronchipret has been proven to be a very safe medicine, it is not expected that it would lead to the development of severe adverse effects in COVID-19 patients. Bronchipret can therefore be recommended as effective and safe supplementary treatments of COVID-19, even more so considering the positive effects shown in vitro. Thus, this randomized study is conducted to assess the effect of Bronchipret on the immune response and recovery in patients with mild COVID-19 by assessing several blood parameters as well as the symptom recovery and improvement in comparison to patients who do not receive Bronchipret. Another aim of this feasibility study is to determine the best possible primary endpoint, i.e. which shows the greatest effect according to Cohen.

DETAILED DESCRIPTION:
Although intensive research efforts have been underway worldwide, so far, only few effective treatment against the disease has been brought to the market in Germany. Based on the pathological features and different clinical phases of COVID-19, particularly in patients with moderate to severe COVID- 19, the classes of drugs used are antiviral agents (e.g., remdesivir), inflammation inhibitors/antirheumatic drugs (e.g., dexamethasone), low molecular weight heparins, plasma, and hyperimmune immunoglobulins Bronchipret exhibits multidirectional anti-inflammatory effects as demonstrated in vitro and in vivo studies. Several clinical trials have demonstrated positive effects of Bronchipret, a fixed combination of thyme herb and ivy leaf fluid extracts, on symptom relieve and recovery time in patients with acute bronchitis and cough. There is currently an urgent need for effective and safe treatments of COVID- 19 and the cytokine storm that is responsible for the development of Acute Respiratory Distress Syndrome (ARDS).

As Bronchipret has been proven to be a very safe medicine, it is not expected that it would lead to the development of severe adverse effects in COVID-19 patients. Bronchipret can therefore be recommended as effective and safe supplementary treatments of COVID-19, even more so considering the positive effects shown in vitro. Thus, this randomized study will be conducted to assess the effect of Bronchipret on the immune response and recovery in patients with mild COVID-19 by assessing several blood parameters as well as the symptom recovery and improvement in comparison to patients who do not receive Bronchipret. Another aim of this feasibility study is to determine the best possible primary endpoint, i.e. which shows the greatest effect according to Cohen.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years and ≤ 75 years

   o If > 50 years, complete COVID-19 vaccination mandatory
2. SARS-CoV-2 infection confirmed by PCR test ≤ 4 days before screening/baseline visit
3. Onset of the earliest symptoms < 7 days before screening/baseline visit
4. Mild COVID-19 with the following symptoms (outpatient management/non hospitalized patients):

   ᴑ Cough and ᴑ At least one other symptom (e.g., sore throat, nasal congestion, headache, nausea, low energy/fatigue, muscle or body ache, shortness of breath, fever, diarrhea, altered sense of smell or taste)
5. Written informed consent obtained prior to the initiation of any protocol-required procedures by the patient
6. Willingness to comply to study procedures and study protocol

Exclusion Criteria:

1. WHO score ≥ 3
2. Other advanced or chronic lung diseases (Chronic obstructive pulmonary disease (COPD), silicosis, bronchial asthma)
3. Unable to take oral medication
4. Body mass index (BMI) > 35 or ≤ 43kg
5. Requirement for oxygen administration
6. Current hospitalization
7. Known hypersensitivity to the active substances ivy, thyme, plants of the aralia family or other labiates (Lamiaceae), birch, mugwort, celery or to any of the excipients
8. Patients with rare hereditary fructose intolerance
9. Inability to monitor body temperature
10. Patients regularly taking immune suppressive medication, nonsteroidal anti-rheumatic drug(s) (NSARs) or steroids (e.g., because of underlying disease)
11. Known significant concomitant diseases or serious and/or uncontrolled diseases that are likely to interfere with the evaluation of the patient's safety and with the study outcome such as stem cell or organ transplantation within the last 5 years, cardiovascular disease, diabetes mellitus, chronic liver disease, chronic kidney disease including dialysis patients, sickle cell anemia or thalassemia, and other forms of immunosuppression (e.g. tumor patients, HIV-infected patients with weakened immune system, iatrogenic immunosuppression) as judged by the study physician according to patient's reports.
12. COVID-19 vaccination planned within study period and/or COVID-19 vaccination within the last 28 days
13. Women pregnant (patient reported at pre-Screening and confirmation via pregnancy test at Screening/baseline) or nursing
14. Males or females of reproductive potential not willing to use effective contraception (defined as PEARL index <1 - e.g. contraceptive pills/intra-uterine devices (IUD))
15. Alcohol, drug or chemical abuse
16. Current participation in another interventional clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in average concentration of immunologic markers | Comparison Baseline to day 7
  concentration of Interleukin 2 (IL-2)
Change in average concentration of immunologic markers - IL4 | Comparison Baseline to day 7
  concentration of Interleukin (IL) 4
Change in average concentration of immunologic markers - Interleukin (IL)-6 | Comparison Baseline to day 7
  concentration of IL-6
Change in average concentration of immunologic markers - IL-8 | Comparison Baseline to day 7
  concentration of IL-8
Change in average concentration of immunologic markers - IL-10 | Comparison Baseline to day 7
  concentration of IL-10
Change in average concentration of immunologic markers - Interferon y | Comparison Baseline to day 7
  concentration of interferon (INF) y
Change in average concentration of immunologic markers- c-reactive protein (CRP) | Comparison Baseline to day 7
  concentration of c-reactive protein (CRP)
Change in average concentration of immunologic markers - IL-1β | Comparison Baseline to day 7
  concentration of IL-1β
Change in average concentration of immunologic markers - Interferon (INF) α | Comparison Baseline to day 7
  concentration of INFα
Change in average concentration of immunologic markers - TNFα | Comparison Baseline to day 7
  concentration of tumor necrosis factor alpha (TNFα)
Change in average number of immunologic markers - neutrophils | Comparison Baseline to day 7
  number of neutrophils
Change in average number of immunologic markers - lymphocytes | Comparison Baseline to day 7
  number of lymphocytes
Change in average number of immunologic markers - monocytes | Comparison Baseline to day 7
  number of monocytes
Change in average number of immunologic markers - eosinophils | Comparison Baseline to day 7
  number of eosinophils
Change in average number of immunologic markers - basophils | Comparison Baseline to day 7
  number of basophils
Change in average number of immunologic markers - platelets | Comparison Baseline to day 7
  number of platelets

SECONDARY OUTCOMES:
Concentration of blood parameters and change to BL - IL2 | Day 4
  percentage of change of concentration of IL-2
Concentration of blood parameters and change to BL | Day 4
  absolute change of concentration of IL-2
Concentration of blood parameters and change to BL (percentage): IL2 | Day 7
  percentage of change of concentration of IL-2
Concentration of blood parameters and change to BL (absolute change): IL2 | Day 7
  absolute change of concentration of IL-2
Concentration of blood parameters and change to BL (absolute change): IL2 | Day 14
  absolute change of concentration of IL-2
Concentration of blood parameters and change to BL (percentage): IL2 | Day 14
  percentage of change of concentration of IL-2
Concentration of blood parameters and change to BL (percentage) IL4 | Day 4
  percentage of change of concentration of IL-4
Concentration of blood parameters and change to BL (absolute change): IL4 | Day 7
  absolute change of concentration of IL-4
Concentration of blood parameters and change to BL (percentage) IL4 | Day 7
  percentage of change of concentration of IL-4
Concentration of blood parameters and change to BL (absolute change) IL4 | Day 14
  absolute change of concentration of IL-4
Concentration of blood parameters and change to BL (percentage) IL4 | Day 14
  percentage of change of concentration of IL-4
Concentration of blood parameters and change to BL (absolute change) IL6 | Day 4
  absolute change of concentration of IL-6
Concentration of blood parameters and change to BL (percentage) IL6 | Day 4
  percentage of change of concentration of IL-6
Concentration of blood parameters and change to BL (absolute change) IL6 | Day 7
  absolute change of concentration of IL-6
Concentration of blood parameters and change to BL (percentage) IL6 | Day 7
  percentage of change of concentration of IL-6
Concentration of blood parameters and change to BL (percentage) IL6 | Day 14
  percentage of change of concentration of IL-6
Concentration of blood parameters and change to BL (absolute change) IL6 | Day 14
  absolute change of concentration of IL-6
Concentration of blood parameters and change to BL (percentage) IL8 | Day 4
  percentage of change of concentration of IL-8
Concentration of blood parameters and change to BL (absolute change) IL8 | Day 4
  absolute change of concentration of IL-8
Concentration of blood parameters and change to BL (percentage): | Day 7
  percentage of change of concentration of IL-8
Concentration of blood parameters and change to BL (absolute change): | Day 7
  absolute change of concentration of IL-8
Concentration of blood parameters and change to BL (percentage): | Day 14
  percentage of change of concentration of IL-8
Concentration of blood parameters and change to BL (absolute change IL8): | Day 14
  absolute change of concentration of IL-8
Concentration of blood parameters and change to BL (absolute change IL10): | Day 4
  absolute change of concentration of IL-10
Concentration of blood parameters and change to BL (IL10 percentage): | Day 4
  percentage of change of concentration of IL-10
Concentration of blood parameters and change to BL (absolute change IL10): | Day 7
  absolute change of concentration of IL-10
Concentration of blood parameters and change to BL (percentage): IL10 | Day 7
  percentage of change of concentration of IL-10
Concentration of blood parameters and change to BL (absolute change IL10): | Day 14
  absolute change of concentration of IL-10
Concentration of blood parameters and change to BL (percentage): IL10 | Day 14
  percentage of change of concentration of IL-10
Concentration of blood parameters and change to BL (INFy percentage): | Day 4
  percentage of change of concentration of INFy
Concentration of blood parameters and change to BL (absolute change INFy): | Day 4
  absolute change of concentration of INFy
Concentration of blood parameters and change to BL (percentage): INFy | Day 7
  percentage of change of concentration of INFy
Concentration of blood parameters and change to BL (absolute change): INFy | Day 7
  absolute change of concentration of INFy
Concentration of blood parameters and change to BL (percentage): INFy | Day 14
  percentage of change of concentration of INFy
Concentration of blood parameters and change to BL (absolute change): INFy | Day 14
  absolute change of concentration of INFy
Concentration of blood parameters and change to BL (absolute change): CRP | Day 4
  absolute change of concentration of CRP
Concentration of blood parameters and change to BL (percentage): CRP | Day 4
  percentage of change of concentration of CRP
Concentration of blood parameters and change to BL (absolute change): CRP | Day 7
  absolute change of concentration of CRP
Concentration of blood parameters and change to BL (percentage): CRP | Day 7
  percentage of change of concentration of CRP
Concentration of blood parameters and change to BL (absolute change): CRP | Day 14
  absolute change of concentration of CRP
Concentration of blood parameters and change to BL (percentage): CRP | Day 14
  percentage of change of concentration of CRP
Concentration of blood parameters and change to BL (percentage): IL-1β | Day 4
  percentage of change of concentration of IL-1β
Concentration of blood parameters and change to BL (absolute change): IL-1β | Day 4
  absolute change of concentration of IL-1β
Concentration of blood parameters and change to BL (percentage): IL-1β | Day 7
  percentage of change of concentration of IL-1β
Concentration of blood parameters and change to BL (absolute change): IL-1β | Day 7
  absolute change of concentration of IL-1β
Concentration of blood parameters and change to BL (percentage): IL-1β | Day 14
  percentage of change of concentration of IL-1β
Concentration of blood parameters and change to BL (absolute change): IL-1β | Day 14
  absolute change of concentration of IL-1β
Concentration of blood parameters and change to BL (absolute change): INFα | Day 4
  absolute change of concentration of INFα
Concentration of blood parameters and change to BL (percentage): INFα | Day 4
  percentage of change of concentration of INFα
Concentration of blood parameters and change to BL (absolute change):INFα | Day 7
  absolute change of concentration of INFα
Concentration of blood parameters and change to BL (percentage): INFα | Day 7
  percentage of change of concentration of INFα
Concentration of blood parameters and change to BL (percentage): INFα | Day 14
  percentage of change of concentration of INFα
Concentration of blood parameters and change to BL (absolute change): INFα | Day 14
  absolute change of concentration of INFα
Concentration of blood parameters and change to BL (absolute change): TNFα, | Day 4
  absolute change of concentration of TNFα,
Concentration of blood parameters and change to BL (percentage): TNFα, | Day 4
  percentage of change of concentration of TNFα,
Concentration of blood parameters and change to BL (absolute change): TNFα, | Day 7
  absolute change of concentration of TNFα,
Concentration of blood parameters and change to BL (percentage): TNFα, | Day 7
  percentage of concentration of TNFα,
Concentration of blood parameters and change to BL (absolute change): TNFα, | Day 14
  absolute change of concentration of TNFα,
Concentration of blood parameters and change to BL (percentage): TNFα, | Day 14
  percentage of change of concentration of TNFα,
Concentration of blood parameters and change to BL (percentage): neutrophils | Day 4
  percentage change of neutrophils
Concentration of blood parameters and change to BL (absolute change): neutrophils | Day 4
  absolute change of neutrophils number
Concentration of blood parameters and change to BL (percentage): neutrophils | Day 7
  percentage change of neutrophils
Concentration of blood parameters and change to BL (absolute change): neutrophils | Day 7
  absolute change of neutrophils number
Concentration of blood parameters and change to BL (percentage): neutrophils | Day 14
  percentage change of neutrophils
Concentration of blood parameters and change to BL (absolute change): neutrophils | Day 14
  absolute change of neutrophils number
Concentration of blood parameters and change to BL (absolute change): lymphocytes | Day 4
  absolute change of lymphocytes number
Concentration of blood parameters and change to BL (percentage): lymphocytes | Day 4
  percentage change of lymphocytes
Concentration of blood parameters and change to BL (absolute change): lymphocytes | Day 7
  absolute change of lymphocytes number
Concentration of blood parameters and change to BL (percentage): lymphocytes | Day 7
  percentage change of lymphocytes
Concentration of blood parameters and change to BL (absolute change): lymphocytes | Day 14
  absolute change of lymphocytes number
Concentration of blood parameters and change to BL (percentage): lymphocytes | Day 14
  percentage change of lymphocytes
Concentration of blood parameters and change to BL (percentage): monocytes | Day 4
  percentage change of monocytes
Concentration of blood parameters and change to BL (absolute change): monocytes | Day 4
  absolute change of monocytes number
Concentration of blood parameters and change to BL (percentage): monocytes | Day 7
  percentage change of monocytes
Concentration of blood parameters and change to BL (absolute change): monocytes | Day 7
  absolute change of monocytes number
Concentration of blood parameters and change to BL (percentage): monocytes | Day 14
  percentage of change of monocytes
Concentration of blood parameters and change to BL (absolute change): monocytes | Day 14
  absolute change of monocytes number
Concentration of blood parameters and change to BL (absolute change): eosinophils | Day 4
  absolute change of eosinophils number
Concentration of blood parameters and change to BL (percentage): eosinophils | Day 4
  percentage of change of eosinophils
Concentration of blood parameters and change to BL (percentage): eosinophils | Day 7
  percentage of change of eosinophils
Concentration of blood parameters and change to BL (absolute change): eosinophils | Day 7
  absolute change of eosinophils number
Concentration of blood parameters and change to BL (percentage): eosinophils | Day 14
  percentage of change of eosinophils
Concentration of blood parameters and change to BL (absolute change): eosinophils | Day 14
  absolute change of eosinophils number
Concentration of blood parameters and change to BL (percentage): | Day 4
  percentage of change of basophils number
Concentration of blood parameters and change to BL (absolute change): | Day 4
  absolute change of basophils number
Concentration of blood parameters and change to BL (absolute change): | Day 7
  absolute change of basophils number
Concentration of blood parameters and change to BL (percentage): | Day 7
  percentage of change of basophils
Concentration of blood parameters and change to BL (absolute change): | Day 14
  absolute change of basophils number
Concentration of blood parameters and change to BL (percentage): | Day 14
  percentage of change of basophils
Concentration of blood parameters and change to BL (percentage): | Day 4
  percentage of change of platelets
Concentration of blood parameters and change to BL (absolute change): | Day 4
  absolute change of platelet number
Concentration of blood parameters and change to BL (percentage): | Day 7
  percentage of change of platelets
Concentration of blood parameters and change to BL (absolute change): | Day 7
  absolute change of platelet number
Concentration of blood parameters and change to BL (percentage): | Day 14
  percentage of change of platelets
Concentration of blood parameters and change to BL (absolute change): | Day 14
  absolute change of platelet number
Concentration of blood parameters and change to BL (percentage): | Day 4
  percentage of change of lactate dehydrogenase (LDH)
Concentration of blood parameters and change to BL (absolute change): | Day 4
  absolute change of lactate dehydrogenase (LDH)
Concentration of blood parameters and change to BL (absolute change): | Day 7
  absolute change of LDH
Concentration of blood parameters and change to BL (percentage): | Day 7
  percentage of change of LDH
Concentration of blood parameters and change to BL (absolute change): | Day 14
  absolute change of LDH
Concentration of blood parameters and change to BL (percentage): | Day 14
  percentage of change of LDH
Concentration of blood parameters and change to BL (percentage): | Day 4
  percentage of change of ferritin
Concentration of blood parameters and change to BL (absolute change): | Day 4
  absolute change of ferritin
Concentration of blood parameters and change to BL (percentage): | Day 7
  percentage of change of ferritin
Concentration of blood parameters and change to BL (absolute change): | Day 7
  absolute change of ferritin
Concentration of blood parameters and change to BL (percentage): | Day 14
  percentage of change of ferritin
Concentration of blood parameters and change to BL (absolute change): | Day 14
  absolute change of ferritin
Concentration of blood parameters and change to BL (absolute change): | Day 4
  absolute change of haemoglobin
Concentration of blood parameters and change to BL (percentage): | Day 4
  percentage of change of haemoglobin
Concentration of blood parameters and change to BL (absolute change): | Day 7
  absolute change of haemoglobin
Concentration of blood parameters and change to BL (percentage): | Day 7
  percentage of change of haemoglobin
Concentration of blood parameters and change to BL (absolute change): | Day 14
  absolute change of haemoglobin
Concentration of blood parameters and change to BL (percentage): | Day 14
  percentage of change of haemoglobin
Concentration of blood parameters and change to BL (absolute change): | Day 4
  absolute change of alanine aminotransferase (ALT)
Concentration of blood parameters and change to BL (percentage): | Day 4
  percentage of change of alanine aminotransferase (ALT)
Concentration of blood parameters and change to BL (absolute change): | Day 7
  absolute change of alanine aminotransferase (ALT)
Concentration of blood parameters and change to BL (percentage): | Day 7
  percentage of change of alanine aminotransferase (ALT)
Concentration of blood parameters and change to BL (percentage): | Day 14
  percentage of change of alanine aminotransferase (ALT)
Concentration of blood parameters and change to BL (absolute change): | Day 14
  absolute change of alanine aminotransferase (ALT)
Concentration of blood parameters and change to BL (absolute change): | Day 4
  absolute change of Aspartate aminotransferase (AST)
Concentration of blood parameters and change to BL (absolute change): | Day 7
  absolute change of Aspartate aminotransferase (AST)
Concentration of blood parameters and change to BL (percentage): | Day 7
  percentage of change of Aspartate aminotransferase (AST)
Concentration of blood parameters and change to BL (absolute change): | Day 14
  absolute change of Aspartate aminotransferase (AST)
Concentration of blood parameters and change to BL (percentage): | Day 14
  percentage of change of Aspartate aminotransferase (AST)
Concentration of blood parameters and change to BL (percentage): | Day 4
  percentage of change of activated partial thromboplastin time
Concentration of blood parameters and change to BL (absolute change): | Day 4
  absolute change of activated partial thromboplastin time
Concentration of blood parameters and change to BL (absolute change): | Day 7
  absolute change of activated partial thromboplastin time
Concentration of blood parameters and change to BL (percentage): | Day 7
  percentage of change of activated partial thromboplastin time
Concentration of blood parameters and change to BL (percentage): | Day 14
  percentage of change of activated partial thromboplastin time
Concentration of blood parameters and change to BL (absolute change): | Day 14
  absolute change of activated partial thromboplastin time
Concentration of blood parameters and change to BL (absolute change): | Day 4
  absolute change of prothrombin Z
Concentration of blood parameters and change to BL (percentage): | Day 4
  percentage of change of prothrombin Z
Concentration of blood parameters and change to BL (absolute change): | Day 7
  absolute change of prothrombin Z
Concentration of blood parameters and change to BL (percentage): | Day 7
  percentage of change of prothrombin Z
Concentration of blood parameters and change to BL (absolute change): | Day 14
  absolute change of prothrombin Z
Concentration of blood parameters and change to BL (percentage): | Day 14
  percentage of change of prothrombin Z
Concentration of blood parameters and change to BL (percentage): | Day 4
  percentage of change of fibrinogen
Concentration of blood parameters and change to BL (absolute change): | Day 4
  absolute change of fibrinogen
Concentration of blood parameters and change to BL (percentage): | Day 7
  percentage of change of fibrinogen
Concentration of blood parameters and change to BL (absolute change): | Day 7
  absolute change of fibrinogen
Concentration of blood parameters and change to BL (percentage): | Day 14
  percentage of change of fibrinogen
Concentration of blood parameters and change to BL (absolute change): | Day 14
  absolute change of fibrinogen
Concentration of blood parameters and change to BL (absolute change): | Day 4
  absolute change of d-dimeric
Concentration of blood parameters and change to BL (percentage): | Day 4
  percentage of change of d-dimeric
Concentration of blood parameters and change to BL (absolute change): | Day 7
  absolute change of d-dimeric
Concentration of blood parameters and change to BL (percentage): | Day 7
  percentage of change of d-dimeric
Concentration of blood parameters and change to BL (absolute change): | Day 14
  absolute change of d-dimeric
Concentration of blood parameters and change to BL (percentage): | Day 14
  percentage of change of d-dimeric
Concentration of blood parameters and change to BL (percentage): | Day 4
  percentage of change of fibrin-degranulation products
Concentration of blood parameters and change to BL (absolute change): | Day 4
  absolute change of fibrin-degranulation products
Concentration of blood parameters and change to BL (percentage): | Day 7
  percentage of change of fibrin-degranulation products
Concentration of blood parameters and change to BL (absolute change): | Day 7
  absolute change of fibrin-degranulation products
Concentration of blood parameters and change to BL (percentage): | Day 14
  percentage of change of fibrin-degranulation products
Concentration of blood parameters and change to BL (absolute change): | Day 14
  absolute change of fibrin-degranulation products
Concentration of blood parameters and change to BL (absolute change): | Day 4
  absolute change of anti-thrombin III activity
Concentration of blood parameters and change to BL (percentage): | Day 4
  percentage of change of anti-thrombin III activity
Concentration of blood parameters and change to BL (absolute change): | Day 7
  absolute change of anti-thrombin III activity
Concentration of blood parameters and change to BL (percentage): | Day 7
  percentage of change of anti-thrombin III activity
Concentration of blood parameters and change to BL (absolute change): | Day 14
  absolute change of anti-thrombin III activity
Concentration of blood parameters and change to BL (percentage): | Day 14
  percentage of change of anti-thrombin III activity
Concentration of blood parameters and change to BL (percentage): | Day 4
  percentage of change of Immunglobulin M (IgM)
Concentration of blood parameters and change to BL (absolute change): | Day 4
  absolute change of Immunglobulin M (IgM)
Concentration of blood parameters and change to BL (percentage): | Day 7
  percentage of change of Immunglobulin M (IgM)
Concentration of blood parameters and change to BL (absolute change): | Day 7
  absolute change of Immunglobulin M (IgM)
Concentration of blood parameters and change to BL (percentage): | Day 14
  percentage of change of Immunglobulin M (IgM)
Concentration of blood parameters and change to BL (absolute change): | Day 14
  absolute change of Immunglobulin M (IgM)
Concentration of blood parameters and change to BL (absolute change): | Day 4
  absolute change of Immunglobulin G (IgG)
Concentration of blood parameters and change to BL (percentage): | Day 4
  percentage of change of Immunglobulin G (IgG)
Concentration of blood parameters and change to BL (absolute change): | Day 7
  absolute change of Immunglobulin G (IgG)
Concentration of blood parameters and change to BL (percentage): | Day 7
  percentage of change of Immunglobulin G (IgG)
Concentration of blood parameters and change to BL (absolute change): | Day 14
  absolute change of Immunglobulin G (IgG)
Concentration of blood parameters and change to BL (percentage): | Day 14
  percentage of change of Immunglobulin G (IgG)
Concentration of blood parameters and change to BL (percentage): | Day 4
  percentage of change of Creatinin
Concentration of blood parameters and change to BL (absolute change): | Day 4
  absolute change of Creatinin
Concentration of blood parameters and change to BL (percentage): | Day 7
  percentage of change of Creatinin
Concentration of blood parameters and change to BL (absolute change): | Day 7
  absolute change of Creatinin
Concentration of blood parameters and change to BL (percentage): | Day 14
  percentage of change of Creatinin
Concentration of blood parameters and change to BL (absolute change): | Day 14
  absolute change of Creatinin
Neutrophil to lymphocyte ratio | Day 4
  Neutrophil to lymphocyte number ratio
Neutrophil to lymphocyte ratio | Day 7
  Neutrophil to lymphocyte number ratio
Neutrophil to lymphocyte ratio | Day 14
  Neutrophil to lymphocyte number ratio
IL-6/IL-10 ratio | Day 4
  IL-6/IL-10 concentration ratio
IL-6/IL-10 ratio | Day 7
  IL-6/IL-10 concentration ratio
IL-6/IL-10 ratio | Day 14
  IL-6/IL-10 concentration ratio
IL-6/INFy ratio | Day 14
  IL-6/INFy concentration ratio
IL-6/INFy ratio | Day 7
  IL-6/INFy concentration ratio
IL-6/INFy ratio | Day 4
  IL-6/INFy concentration ratio
Assessment of symptom improvement/worsening | Day 4
  FDA (Federal drug agency) recommended symptom questionnaire - higher scores describe worse symptoms, scoring 0 to 3 (question 1 to 12) and 0 to 2 (question 13 and 14)
Assessment of symptom improvement/worsening | Day 7
  FDA (Federal drug agency) recommended symptom questionnaire - higher scores describe worse symptoms, scoring 0 to 3 (question 1 to 12) and 0 to 2 (question 13 and 14)
Assessment of symptom improvement/worsening | Day 14
  FDA (Federal drug agency) recommended symptom questionnaire - higher scores describe worse symptoms, scoring 0 to 3 (question 1 to 12) and 0 to 2 (question 13 and 14)
Assessment of symptom improvement/worsening | Day 28
  FDA (Federal drug agency) recommended symptom questionnaire - higher scores describe worse symptoms, scoring 0 to 3 (question 1 to 12) and 0 to 2 (question 13 and 14)
Assessment of number of symptoms | Day 4
  FDA (Federal drug agency) recommended symptom questionnaire - higher scores describe worse symptoms, scoring 0 to 3 (question 1 to 12) and 0 to 2 (question 13 and 14)
Assessment of number of symptoms | Day 7
  FDA (Federal drug agency) recommended symptom questionnaire - higher scores describe worse symptoms, scoring 0 to 3 (question 1 to 12) and 0 to 2 (question 13 and 14)
Assessment of number of symptoms | Day 14
  FDA (Federal drug agency) recommended symptom questionnaire - higher scores describe worse symptoms, scoring 0 to 3 (question 1 to 12) and 0 to 2 (question 13 and 14)
Assessment of number of symptoms | Day 28
  FDA (Federal drug agency) recommended symptom questionnaire - higher scores describe worse symptoms, scoring 0 to 3 (question 1 to 12) and 0 to 2 (question 13 and 14)
Assessment of symptom distribution | Day 4
  FDA (Federal drug agency) recommended symptom questionnaire - higher scores describe worse symptoms, scoring 0 to 3 (question 1 to 12) and 0 to 2 (question 13 and 14)
Assessment of symptom distribution | Day 7
  FDA (Federal drug agency) recommended symptom questionnaire - higher scores describe worse symptoms, scoring 0 to 3 (question 1 to 12) and 0 to 2 (question 13 and 14)
Assessment of symptom distribution | Day 14
  FDA (Federal drug agency) recommended symptom questionnaire - higher scores describe worse symptoms, scoring 0 to 3 (question 1 to 12) and 0 to 2 (question 13 and 14)
Assessment of symptom distribution | Day 28
  FDA (Federal drug agency) recommended symptom questionnaire - higher scores describe worse symptoms, scoring 0 to 3 (question 1 to 12) and 0 to 2 (question 13 and 14)
Assessment of defervescence | Day 28
  Time to defervescence in days
Assessment of defervescence - number of patients | Day 28
  Number of patients who achieved defervescence
Assessment of defervescence - portion of patients | Day 28
  Proportion of patients who achieved defervescence
Assessment of defervescence | Day 4
  Absolute temperature values and change to BL
Assessment of defervescence | Day 7
  Absolute temperature values and change to BL
Assessment of defervescence | Day 14
  Absolute temperature values and change to BL
Assessment of defervescence | Day 28
  Absolute temperature values and change to BL
Assessment of improvement or absence of coughing | Day 28
  Time to cough reported as mild oder non existent in days
Assessment of improvement or absence of coughing | Day 28
  Time to non-existent coughing for all patients in days
Assessment of improvement or absence of coughing - proportion of patients | Day 28
  proportion of patients with moderate or severe cough at BL who achieved cough reported as mild or none existent
Assessment of improvement or absence of coughing - number of patients | Day 28
  Number of patients with moderate or severe cough at BL who achieved cough reported as mild or none existent
Assessment of improvement or absence of coughing | Day 28
  proportion of patients who achieved cough reported as none existent
Assessment of intensity and distribution of most bothersome symptom | Day 28
  Intensity of most bothersome symptom assessment done by visual analogue scale (VAS) and change to Baseline - score 0 to 10 cm, higher values describe higher intensity
Assessment of intensity and distribution of most bothersome symptom | Day 28
  Most bothersome symptom distribution (i.e.,number and percentage of patients with each symptom) (the most bothersome symptom will be defined by the patient at BL) assessment done by visual analogue scale (VAS) - score 0 to 10 cm, higher values describe higher intensity
Proportion of patients who return to usual health | Day 28
  proportion of patients who return to usual health
Number of patients who return to usual health | Day 28
  Number of patients who return to usual health
proportion of patients who return to usual activity | Day 28
  proportion of patients who return to usual activity
Requirement of hospitalisation or oxygen supplementation | Day 28
  Number of patients requiring hospitalisation or oxygen supplementation (patient reported)
Requirement of hospitalisation or oxygen supplementation | Day 28
  proportion of patients requiring hospitalisation or oxygen supplementation (patient reported)
Disease progression/improvement | Day 4
  Number of patients with improved or progressed disease state (according to world health organisation (WHO) scale) - Score 0 - 10, higher score described more progressed state
Disease progression/improvement | Day 4
  proportion of patients with improved or progressed disease state (according to world health organisation (WHO) scale) - Score 0 - 10, higher score described more progressed state
Disease progression/improvement | Day 7
  Number of patients with improved or progressed disease state (according to world health organisation (WHO) scale) Score 0 - 10, higher score described more progressed state
Disease progression/improvement | Day 7
  proportion of patients with improved or progressed disease state (according to world health organisation (WHO) scale) Score 0 - 10, higher score described more progressed state
Disease progression/improvement | Day 14
  Number of patients with improved or progressed disease state (according to world health organisation (WHO) scale) Score 0 - 10, higher score described more progressed state
Disease progression/improvement | Day 14
  proportion of patients with improved or progressed disease state (according to world health organisation (WHO) scale), Score 0 - 10, higher score described more progressed state
Disease progression/improvement | Day 28
  Number of patients with improved or progressed disease state (according to world health organisation (WHO) scale) Score 0 - 10, higher score described more progressed state
Disease progression/improvement | Day 28
  proportion of patients with improved or progressed disease state (according to world health organisation (WHO) scale) Score 0 - 10, higher score described more progressed state
Disease progression/improvement | Day 4
  Number of patients with each WHO score Score 0 - 10, higher score described more progressed state
Disease progression/improvement | Day 4
  proportion of patients with each WHO score Score 0 - 10, higher score described more progressed state
Disease progression/improvement | Day 7
  Number of patients with each WHO score Score 0 - 10, higher score described more progressed state
Disease progression/improvement | Day 7
  proportion of patients with each WHO score Score 0 - 10, higher score described more progressed state
Disease progression/improvement | Day 14
  Number of patients with each WHO score Score 0 - 10, higher score described more progressed state
Disease progression/improvement | Day 14
  proportion of patients with each WHO score Score 0 - 10, higher score described more progressed state
Disease progression/improvement | Day 28
  Number of patients with each WHO score Score 0 - 10, higher score described more progressed state
Disease progression/improvement | Day 28
  proportion of patients with each WHO score Score 0 - 10, higher score described more progressed state
Disease progression/improvement | Day 4
  WHO score and change to BL Score 0 - 10, higher score described more progressed state
Disease progression/improvement | Day 7
  WHO score and change to BL Score 0 - 10, higher score described more progressed state
Disease progression/improvement | Day 14
  WHO score and change to BL Score 0 - 10, higher score described more progressed state
Disease progression/improvement | Day 28
  WHO score and change to BL Score 0 - 10, higher score described more progressed state
Disease progression/improvement | Day 4
  Number of patients in each disease severity state according to WHO score Score 0 - 10, higher score described more progressed state
Disease progression/improvement | Day 4
  proportion of patients in each disease severity state according to WHO score Score 0 - 10, higher score described more progressed state
Disease progression/improvement | Day 7
  Number of patients in each disease severity state according to WHO score Score 0 - 10, higher score described more progressed state
Disease progression/improvement | Day 7
  proportion of patients in each disease severity state according to WHO score Score 0 - 10, higher score described more progressed state
Disease progression/improvement | Day 14
  proportion of patients in each disease severity state according to WHO score Score 0 - 10, higher score described more progressed state
Disease progression/improvement | Day 14
  Number of patients in each disease severity state according to WHO score Score 0 - 10, higher score described more progressed state
Disease progression/improvement | Day 28
  proportion of patients in each disease severity state according to WHO score Score 0 - 10, higher score described more progressed state
Disease progression/improvement | Day 28
  Number of patients in each disease severity state according to WHO score Score 0 - 10, higher score described more progressed state
Assessment of oxygen saturation | Day 4
  Oxygen saturation measured by finger clip and change to BL
Assessment of oxygen saturation | Day 7
  Oxygen saturation measured by finger clip and change to BL
Assessment of oxygen saturation | Day 14
  Oxygen saturation measured by finger clip and change to BL
Assessment of oxygen saturation | Day 28
  Oxygen saturation measured by finger clip and change to BL
Assessment of intake of concomitant medication | Day 14
  Type and average daily dose of concomitant medication and total dose of paracetamol
Assessment of intake of concomitant medication | Day 4
  Average days of additional intake of concomitant medication paracetamol
Assessment of intake of concomitant medication | Day 7
  Average days of additional intake of concomitant medication paracetamol
Assessment of intake of concomitant medication | Day 14
  Average days of additional intake of concomitant medication paracetamol
Assessment of intake of concomitant medication | Day 28
  Average days of additional intake of concomitant medication paracetamol
Assessment of intake of concomitant medication | Day 14
  Number of patients with a reduction in concomitant medication intake
Assessment of intake of concomitant medication | Day 14
  proportion of patients with a reduction in concomitant medication intake
Number of patients with hyposmia or anosmia | Day 4
  Number of patients with hyposmia or anosmia
proportion of patients with hyposmia or anosmia | Day 4
  proportion of patients with hyposmia or anosmia
Number of patients with hyposmia or anosmia | Day 7
  Number of patients with hyposmia or anosmia
proportion of patients with hyposmia or anosmia | Day 7
  proportion of patients with hyposmia or anosmia
Number of patients with hyposmia or anosmia | Day 14
  Number of patients with hyposmia or anosmia
proportion of patients with hyposmia or anosmia | Day 14
  proportion of patients with hyposmia or anosmia
Number of patients with hyposmia or anosmia | Day 28
  Number of patients with hyposmia or anosmia
proportion of patients with hyposmia or anosmia | Day 28
  proportion of patients with hyposmia or anosmia
Number of patients with fever | Day 4
  Number of patients with fever
proportion of patients with fever | Day 4
  proportion of patients with fever
Number of patients with fever | Day 7
  Number of patients with fever
proportion of patients with fever | Day 7
  proportion of patients with fever
Number of patients with fever | Day 14
  Number of patients with fever
proportion of patients with fever | Day 14
  proportion of patients with fever
Number of patients with fever | Day 28
  Number of patients with fever
proportion of patients with fever | Day 28
  proportion of patients with fever
Number of patients with COVID-19 vaccination | Day 4
  Number of patients with COVID-19 vaccination
proportions of patients with COVID-19 vaccination | Day 4
  proportions of patients with COVID-19 vaccination
Number of patients with COVID-19 vaccination | Day 7
  Number of patients with COVID-19 vaccination
proportions of patients with COVID-19 vaccination | Day 7
  proportions of patients with COVID-19 vaccination
Number of patients with COVID-19 vaccination | Day 14
  Number of patients with COVID-19 vaccination
proportions of patients with COVID-19 vaccination | Day 14
  proportions of patients with COVID-19 vaccination
Number of patients with COVID-19 vaccination | Day 28
  Number of patients with COVID-19 vaccination
proportions of patients with COVID-19 vaccination | Day 28
  proportions of patients with COVID-19 vaccination
Number of recovered COVID-19 patients | Day 4
  Number of recovered COVID-19 patients
proportion of recovered COVID-19 patients | Day 4
  proportion of recovered COVID-19 patients
Number of recovered COVID-19 patients | Day 7
  Number of recovered COVID-19 patients
proportion of recovered COVID-19 patients | Day 7
  proportion of recovered COVID-19 patients
Number of recovered COVID-19 patients | Day 14
  Number of recovered COVID-19 patients
proportion of recovered COVID-19 patients | Day 14
  proportion of recovered COVID-19 patients
Number of recovered COVID-19 patients | Day 28
  Number of recovered COVID-19 patients
proportion of recovered COVID-19 patients | Day 28
  proportion of recovered COVID-19 patients
Assessment of severe acute respiratory syndrome (SARS)- Corona virus (CoV) -2 negativity | Day 4
  Assessment of SARS-CoV-2 negativity measured by polymerase chain reaction (PCR) test)
Assessment of SARS-CoV-2 negativity | Day 7
  Assessment of SARS-CoV-2 negativity measured by polymerase chain reaction (PCR) test)
Assessment of SARS-CoV-2 negativity | Day 14
  Assessment of SARS-CoV-2 negativity measured by polymerase chain reaction (PCR) test)
Assessment of SARS-CoV-2 negativity | Day 28
  Assessment of SARS-CoV-2 negativity measured by polymerase chain reaction (PCR) test)
Assessment of compliance | Day 4
  Compliance to investigational medicinal product (IMP) by dose taken and as documented in patient diary
Assessment of compliance | Day 7
  Compliance to IMP by dose taken and as documented in patient diary
Assessment of compliance | Day 14
  Compliance to IMP by dose taken and as documented in patient diary
Number of adverse events (AE) | through study completion, average 28 days
  Number of adverse events (AE)
Number of serious adverse events (SAE) | through study completion, average 28 days
  Number of serious adverse events (SAE)
Type and severity of adverse events | through study completion, average 28 days
  Type and severity of adverse events
Type and severity of serious adverse events | through study completion, average 28 days
  Type and severity of serious adverse events
Seriousness and relatedness of AEs | through study completion, average 28 days
  Seriousness and relatedness of AEs
Seriousness and relatedness of SAEs | through study completion, average 28 days
  Seriousness and relatedness of SAEs

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Schaefer, MD, Principal Investigator — Fraunhofer ITMP
Locations (1):
- Fraunhofer ITMP - early clinical development, Frankfurt, Hessia, Germany

IPD SHARING:
Plan to Share IPD: No